CLINICAL TRIAL: NCT04858919
Title: Transrectal Ultrasound and 3D Transabdominal Ultrasound in Comparison to Vaginoscopy in Virgins With Suspected Genital Tract Lesions
Brief Title: Transrectal and 3D Transabdominal Ultrasound Compared to Vaginoscopy in Diagnosing Virgins With Genital Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: vaginoscope
Record Dates: First submitted 2021-04-13; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Virginity; Genital Diseases, Female; Diagnoses Disease
MeSH Terms: conditions — Sexual Abstinence; Genital Diseases, Female

STUDY DESIGN:
Intervention Model Description: A diagnostic test accuracy study that will be conducted at Ain-Shams University Maternity Hospital ,the patients will be recruited from women admitted from gynecologic clinic or from emergency room and from patients following up in outpatient clinic patients will be recruited to this study All Patients recruited must have suspected uterine, cervical or vaginal lesion by history, examination and Pelvic ultrasound
Masking Description: The sonographers will be blinded to all images obtained from the initial pelvic ultrasound and from the images obtained by the alternative sonographic modality. Also All sonographic images will be concealed from the physicians performing the vaginoscopy procedure .
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Other): virgins with genital tract lesion
  Interventions: Diagnostic Test: 3D transabdominal ultrasound; Diagnostic Test: transrectal ultrasound; Diagnostic Test: vaginoscopy

INTERVENTIONS:
Diagnostic Test: 3D transabdominal ultrasound — Initially 3D pelvic ultrasound will be performed on all patients. The transabdominal probes used will be those of the ultrasound scanner using a convex probe (multiple frequency 1-6 MHz).
Diagnostic Test: transrectal ultrasound — The vaginal probe will be covered with the customary plastic sheath and richly lubricated with lubricating gel. The probe will then be slowly advanced into the rectum. The transvaginal probes used will be those of the ultrasound scanner using a vaginal probe (multiple frequency 1-8 MHz). The scanning technique will be similar to that of Transvaginal ultrasound.
Diagnostic Test: vaginoscopy — It is the final procedure in the study to reach the accurate diagnosis. A rigid hysteroscope will be used. The sheath has a 5-mm outer diameter, with 2.9 mm rod lens. A high intensity light source and fiberoptic cable will be used to illuminate the uterine cavity. A solution of 0.9% normal saline will be used as the distention medium. The pressure will be kept at 100-120 mmHg using a pressure adjustable cuff system with the aim of maintaining the lowest pressure required to distend the uterine cavity.

SUMMARY:
This study is to compare the feasibility and test performance of different 3D pelvic ultrasound and Transrectal ultrasound in the detection of local lesions in the uterus , cervix and vagina compared to the final diagnosis confirmed by vaginoscopy as a golden standard modality of diagnosis in Virgin Patients

DETAILED DESCRIPTION:
Virginity is a very private issue; saving or losing it is a matter of choice depending on age, ethnicity, religion, or simply personal decision. Post-pubertal teenage girls, religious women such as nuns, and women in some countries tend to be virgin. This situation must be respected by medical professionals. But when a vaginal examination is necessary, virginity might be a limiting factor for the gynecologist in diagnosis and treatment.

Vaginal discharge or bleeding is the symptom most commonly reported by adolescent girls that are referred for gynecologic problems. The most common cause of vaginal discharge at these ages is infection due to a hypo-estrogenized vagina, although other potential causes, such as congenital anomalies of the genitalia, trauma, foreign bodies, sexual abuse, and malignant disease, must also be excluded. With regard to virginity and childbearing possibility in the future, a careful approach is of paramount importance.

Hymenal tissue does not easily tolerate vigorous manipulation and wide movements. When needed, potential hymeneal disruption may be discussed with mature women or with the parents of adolescent girls for the sake of correct diagnosis and treatment; but in general, they are highly resistant to that.

When a reproductive tract examination or transvaginal operation must be arranged for a virgin, the operator faces a challenge and may hesitate to utilize hysteroscopy, which can result in a delayed diagnosis or improper treatment.

The most common indication for hysteroscopy is abnormal vaginal bleeding in virginal patients and has been widely used for uterine cavity examination and management. Although the possibility of hymen preservation is high, virgins are highly resistant to this procedure. This may be due to a belief that the procedure causes disruption of virginity and worries associated with their future partners.

The approach by vaginoscopy and hysteroscopy via a hysteroscope provides a safe and non-traumatic method in assessing the reproductive organs because the scope of the hysteroscope is advanced into the vagina without a speculum or tenaculum. Distension of the vaginal wall by distension medium can in turn provide a clear endoscopic view.

These considerations have made clinicians opt for these procedures in assessing pathologies of the vagina, the surface of the cervix, the cervical canal, and the intrauterine cavity and other developmental anomalies of the sex organs in patients. Furthermore, the entire procedure can be undertaken without disrupting integrity of the hymen, whereas the traditional method requires the use of retractors and, therefore, disrupts this integrity.

Although hysteroscopy can improve diagnosis and thereby improve quality of life, virgins may decline this procedure. Patients with delayed diagnosis and management in some uncommon but serious situations, such as endometrial malignancy, are life-threatening.

So far, only a few reports have discussed the protection of hymen integrity in hysteroscopy, and the physical and psychological impacts of this surgery in virgins are not conclusive .This is an important issue that gynecologists encounter, but which has seldom been discussed. Intravenous sedation is recommended to reduce the patient's anxiety and pain, avoid vasovagal reaction, relax the buttock muscles and reduce the risk of hymenal trauma . Unlike operative hysteroscope, loop electrode cannot be employed in mini-hysteroscope; therefore, for some diseases like submucous leiomyoma or uterine septum, mini-hysteroscopy is not therapeutically beneficial, and this should be explained to the patients in advance. Adequate preoperative counseling is also necessary to emphasize the importance of the procedure and to lessen their anxiety.

In virgin patients when vaginal examination cannot be done ultrasonography is a useful adjunct to inspection of the external genital organs.

Currently there are three accepted and more or less widely used modalities to image the contents of the female pelvis. Transabdominal sonography (TAS) was the first to be used and is still the most widespread.

By using a full urinary bladder as an acoustic window, ovaries, uterus, and superior vagina can be clearly examined using transabdominal (TA) ultrasonography.

Transvaginal sonography provides clear images of the region of interest, provided that the targeted organ is within the focal range of the probe, and that the probe is placed in proximity to the organ in question .

Agenesis of the vagina, a virginal introitus and the fear of introducing infection such as in the case of premature rupture of the membranes are some of the more common situations in which Transvaginal ultrasound is not possible or is relatively contraindicated.

In such cases introducing a commercially available vaginal probe through the anal sphincter into the rectum seems to be a reasonable alternative to image the female pelvic structures within 'reach' of the probe. We present a study to compare TAS and transrectal sonography (TRS) in a group of patients in whom Transvaginal ultrasound was not possible.

Transrectal sonography (TRUS) has been widely used in men as a diagnostic tool for prostate cancer. Its value in the management of disorders of the lower urinary tract in women and as an alternative to intraoperative gynecologic sonography has also been documented . Case reports in the radiological literature attest to the fact that it has been used to guide drainage of inflammatory pelvic collections.

ELIGIBILITY:
Inclusion Criteria:

* Virgins complaining of Abnormal vaginal bleeding, abnormal discharge , pelvic pain
* Virgins with Suspected genital tract lesion by examination
* Virgins with Suspected genital tract lesion by pelvic ultrasound

Exclusion Criteria:

* Sexually Active Patients
* Suspected or documented Pregnancy
* Virgin patients with no suspected uterine, cervical or vaginal lesion by pelvic ultrasound
* Patients unable to communicate effectively

Ages: 5 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of different diagnostic modalities in Virgins. | 1 to 2 hours
  By questionnaire to asses the acceptance of patient to undergo different modalities as 3D pelvic ultrasound, Transrectal ultrasound and vaginoscopy is assessed.
Test performance of different diagnostic modalities in Virgins | 24 hours to 1 week
  diagnostic accuracy of 3D pelvic ultrasound and Transrectal ultrasound in the detection of local lesions in the uterus, cervix and vagina compared to the final diagnosis confirmed by vaginoscopy as a golden standard modality of diagnosis in Virgins.

SECONDARY OUTCOMES:
Patients' satisfaction | 1-2 hours
  Visual Analogue Scale will be used for grading levels of patients' overall satisfaction by giving a range of potential scores (0-10) with a score 0 reflecting greatest satisfaction
patients' pain | 1-2 hours
  Visual Analogue Scale will be used for grading levels of patients' pain by giving a range of potential scores (0-10) with a score 0 reflecting least discomfort

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 6 months after publishing